CLINICAL TRIAL: NCT04700839
Title: The Efficacy of Canagliflozin Versus Metformin in Women With Polycystic Ovary Syndrome: A Randomized, Open Label Trial
Brief Title: SGLT2 Inhibitors in Patients With PCOS
Acronym: PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Director, Principal Investigator, Clinical Professor, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGLT2i PCOS
Record Dates: First submitted 2020-08-05; First posted 2021-01-08 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic ovary syndrome (PCOS);; Insulin resistance (IR); Sodium-glucose co-transporter-2 inhibitors (SGLT-2i); Canagliflozin
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Sodium-Glucose Transporter 2 Inhibitors; Canagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SGLT2 inhibitors group (Experimental): Intervention with SGLT2 inhibitors (100mg/d) for 3 months
  Interventions: Drug: SGLT2 inhibitors
- Metformin group (Active Comparator): Intervention with metformin (1500-2000mg/d) for 3 months
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: SGLT2 inhibitors — Sodium-glucose cotransporters inhibitors (SGLT2i) are novel hypoglycemic drugs with unique hypoglycemic mechanisms, which are completely independent of islet β-cell function or insulin sensitivity. Previous studies have shown that SGLT2i may improve IR by inhibiting glucotoxicity, reducing body weight, reducing inflammation, improving islet β-cell function, and reducing oxidative stress.
  Other Names: Canagliflozin tablets or Glucophage
  Arms: SGLT2 inhibitors group
Drug: Metformin — Metformin is a classic drug for the treatment of polycystic ovary syndrome, which can improve the degree of insulin resistance in PCOS patients.
  Arms: Metformin group

SUMMARY:
Polycystic ovary syndrome (PCOS) is a common endocrine disorder, with a prevalence of 5% to 15% in premenopausal women. Patients with PCOS presents as abnormal menstruation, ovulation disorders and/or hyperandrogenemia, and often accompanied by insulin resistance and other metabolic abnormalities. Metformin has been clarified as an option in patients with PCOS. However, the clinical responses to metformin are limited and different. Sodium glucose co-transporter 2 (SGLT2) inhibitors are novel drugs for the treatment of type 2 diabetes, with weight loss, reducing insulin resistance and cardiovascular benefits. Limited data is available on the efficacy of SGLT2 inhibitors in patients with PCOS.

DETAILED DESCRIPTION:
This clinical study aims to determine the safety and efficacy of canagliflozin vs metformin in Polycystic Ovary Syndrome (PCOS) patients with insulin resistance (IR). Methods: A single center, prospective, randomized open-label study (ratio 1:1), non-inferiority trial was conducted in the department of endocrinology, Shanghai Tenth People's Hospital between July 2019 and April 2021. PCOS women aged 18-45 years with IR were enrolled and randomly assigned to either canagliflozin 100 mg (n = 33) or metformin 1500-2000 mg (n = 35) daily for 12 weeks. The primary outcome was changes in HOMA-IR after 12 weeks treatment. The secondary outcomes included changes in anthropometric, menstrual frequency, sex hormone and metabolic parameters.

ELIGIBILITY:
Inclusion criteria:

* Fmale aged 18- 45;
* Meet Rotterdam criteria;
* Insulin Rsistance

Exclusion Criteria:

* Women who are pregnant or have a pregnancy plan within six months; ·Congenital adrenocortical hyperplasia;
* Hyperprolactinemia;
* Hyperthyroidism or hypothyroidism;
* Abnormal liver function (≥ 3 times of the upper limit of normal range);
* Abnormal renal function (GFR<60ml/min/1.73m2);
* Adrenal or ovarian tumors secreting androgens;
* Used contraceptives, metformin, GLP-1RA, SGLT2I, pioglitazone and contraceptives in the last 3 month.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 3 months
  Homeostatic model assessment insulin resistance index

SECONDARY OUTCOMES:
WHR | 3 months
  Waist/hip Ratio
WC | 3 months
  Waist Circumference (cm）
HC | 3 months
  Hip Circumference（cm）
Menstrual cycles | 3 months
  annual number of menstrual cycles
FBG | 3 months
  fasting blood-glucose in mmol/L
PBG | 3 months
  postprandial blood-glucose in mmol/L
FINS | 3 months
  fasting serum insulin in mU/L
PINS | 3 months
  Postprandial insulin in mU/L
ALT | 3 months
  alanine aminotransferase in U/L
AST | 3 months
  Aspartate aminotransferase in U/L
UA | 3 months
  Uric acid in umol/L
CR | 3 months
  Creatinine in umol/L
LDL-c | 3 months
  low-density lipoprotein cholesterol in mmol/L
HDL-c | 3 months
  high-density lipoprotein cholesterol in mmol/L
TC | 3 months
  Total Cholesterol in mmol/L
TG | 3 months
  Triglyceride in mmol/L
TT | 3 months
  total testosterone in nmol/L
LH | 3 months
  Luteinizing hormone in IU/L
FSH | 3 months
  follicle-stimulating hormone in IU/L）
E2 | 3 months
  Estradiol in pmol/L、PRL(Prolactin in uIU/ml)
PRL | 3 months
  Prolactin in uIU/ml
Metabonomics | 3 months
  the change of Metabonomics after the treatment
Ferriman-Gallwey score | 3 months
  Ferriman-Gallwey score、acne, male pattern baldness
acne score | 3 months
  male pattern baldness
male pattern baldness | 3 months
  male pattern baldness
HOMA- ISI | 3 months
  Homeostatic model assessment insulin sensitivity index
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 3 months
  Adverse events and Safety data in two treatment groups.
BMI | 3 months
  body mass index in kg/m^2
SHBG | 3 months
  sex hormone binding globulin in nmol/L
FT | 3 months
  Free testosterone in pg/ml
DHEAS | 3 months
  Dehydroepiandrosterone Sulfate in ug/dl
AD | 3 months
  Androstenedione in ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Shen Qu, Dr, Study Chair — Shang hai Tenth People's Hospital
Locations (1):
- Shanghai Tenth People' Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Javed Z, Papageorgiou M, Deshmukh H, Rigby AS, Qamar U, Abbas J, Khan AY, Kilpatrick ES, Atkin SL, Sathyapalan T. Effects of empagliflozin on metabolic parameters in polycystic ovary syndrome: A randomized controlled study. Clin Endocrinol (Oxf). 2019 Jun;90(6):805-813. doi: 10.1111/cen.13968. Epub 2019 Apr 2. PMID 30866088
- [Derived] Yan Q, Cai M, Wang N, Wu W, Zhang H, Zhu Y, Luo J, Zhang M, Li J. Circulating Profiles of the Bile Acid Metabolomics in Patients With Polycystic Ovary Syndrome Treated With Metformin or Canagliflozin. Pharmacotherapy. 2025 Dec 16. doi: 10.1002/phar.70092. Online ahead of print. PMID 41401816
- See also: Efficacy of canagliflozin versus metformin in women with polycystic ovary syndrome: A randomized, open-label, noninferiority trial — https://pubmed.ncbi.nlm.nih.gov/34726324/
- See also: Effects of empagliflozin on metabolic parameters in polycystic ovary syndrome: a randomized controlled study — https://pubmed.ncbi.nlm.nih.gov/30866088/